CLINICAL TRIAL: NCT01234337
Title: A Phase III Randomized, Double Blind, Placebo-controlled Trial Comparing Capecitabine Plus Sorafenib Versus Capecitabine Plus Placebo in the Treatment of Locally Advanced or Metastatic HER2-Negative Breast Cancer
Brief Title: Phase III Trial Comparing Capecitabine in Combination With Sorafenib or Placebo in the Treatment of Locally Advanced or Metastatic HER2-Negative Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Onyx Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12444; 2010-018501-10 (EudraCT Number)
Record Dates: First submitted 2010-10-04; First posted 2010-11-04 (Estimated); Results first posted 2015-09-03 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; HER2-neu
MeSH Terms: conditions — Breast Neoplasms | interventions — Sorafenib; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sorafenib (Nexavar, BAY43-9006) + Capecitabine (Experimental): Capecitabine was administered orally at a dose of 1,000 milligram per square meter (mg/m^2) twice daily (12 hours apart) on Days 1 through 14 of each 21-day cycle. Sorafenib was administered orally at a dose of 600 mg (200 mg in the morning, 400 mg in the evening) daily, continuously (that is, Days 1 to 21, inclusive). A treatment cycle consisted of 21 days. If tolerability criteria were met for a subject, capecitabine dose was escalated to 1,250 mg/m^2 twice daily and sorafenib dose to a total daily dose of 800 mg for that subject.
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006); Drug: Capecitabine
- Placebo + Capecitabine (Placebo Comparator): Capecitabine was administered orally at a dose of 1,000 mg/m^2 twice daily (12 hours apart) on Days 1 through 14 of each 21-day cycle. Placebo matching to sorafenib was administered orally, 3 tablets (1 tablet in the morning, 2 tablets in the evening) daily, continuously (that is, Days 1 to 21, inclusive). A treatment cycle consisted of 21 days. If tolerability criteria were met for a subject, capecitabine dose was escalated to 1,250 mg/m^2 twice daily and placebo dose to a total daily dose of 4 tablets (2 tablets twice daily) for that subject.
  Interventions: Drug: Placebo; Drug: Capecitabine

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Capecitabine was administered orally at a dose of 1,000 milligram per square meter (mg/m^2) twice daily (12 hours apart) on Days 1 through 14 of each 21-day cycle. Sorafenib was administered orally at a dose of 600 mg (200 mg in the morning, 400 mg in the evening) daily, continuously (that is, Days 1 to 21, inclusive). A treatment cycle consisted of 21 days. If tolerability criteria were met for a subject, capecitabine dose was escalated to 1,250 mg/m^2 twice daily and sorafenib dose to a total daily dose of 800 mg for that subject.
  Arms: Sorafenib (Nexavar, BAY43-9006) + Capecitabine
Drug: Placebo — Capecitabine was administered orally at a dose of 1,000 mg/m^2 twice daily (12 hours apart) on Days 1 through 14 of each 21-day cycle. Placebo matching to sorafenib was administered orally, 3 tablets (1 tablet in the morning, 2 tablets in the evening) daily, continuously (that is, Days 1 to 21, inclusive). A treatment cycle consisted of 21 days. If tolerability criteria were met for a subject, capecitabine dose was escalated to 1,250 mg/m^2 twice daily and placebo dose to a total daily dose of 4 tablets (2 tablets twice daily) for that subject.
  Arms: Placebo + Capecitabine
Drug: Capecitabine — Capecitabine was administered orally at a dose of 1,000 milligram per square meter (mg/m^2) twice daily (12 hours apart) on Days 1 through 14 of each 21-day cycle.days. If tolerability criteria were met for a subject, capecitabine dose was escalated to 1,250 mg/m^2 twice daily,

SUMMARY:
The objective of this phase-III trial is to compare the efficacy and safety of sorafenib in combination with capecitabine versus capecitabine in combination with placebo in the treatment of subjects with locally advanced or metastatic HER2-negative breast cancer who are resistant to or have failed prior taxane and an anthracycline or for whom further anthracycline therapy is not indicated. After signing consent there can be up to 28 days before starting the treatment during which time a number of tests will be carried out which will include tumor evaluations and medical history. The following tests and evaluations will have to be done within 7 days of the start of treatment,on Day 1 of every cycle and at the end of study: Electrocardiogram, blood tests, patient quality of life questionnaires and a complete physical exam and vital signs. Treatment will be given in 21 day cycles with sorafenib/placebo to be taken every day for 21 days and capecitabine to be taken for the first 14 days. Patients will come in weekly for the first 6 weeks and then on Day1 for every cycle after the first 2 cycles. During the weekly visits the subjects will be check for any side effects and blood draws will happen for the study on Day 1 of each cycle. Subjects will be followed for overall survival.

DETAILED DESCRIPTION:
Research summary (NRES, UK):

Breast cancer is the most commonly diagnosed cancer in women and the leading cause of cancer-related death among women worldwide.

However, despite advances in treatment of the early-stage disease, about 25-40% of patients will develop recurrence or spread to other parts of the body that is largely incurable. The average survival of patients with breast cancer that has spread to other parts of the body (metastasis) is 2 to 3 years after diagnosis, and although a number of treatment options are available, including various chemotherapy agents, no single standard of care exists.

The study drug (Sorafenib) works by inhibiting certain pathways in the body that contribute to tumour growth and the formation of new blood vessels (angiogenesis). Angiogenesis plays an important role in the development, transformation and spread of breast cancer. Capecitabine is an approved chemotherapy drug for patients whose breast cancer has spread to other parts of the body (metastatic) and is not responsive to other classes of chemotherapy drugs.

Data from a Phase IIb clinical study suggests that there is a role for the combination of Sorafenib and Capecitabine to treat locally advanced or metastatic breast cancer.

Patients in this confirmatory Phase III study will be randomly assigned to receive either:

* Capecitabine + Sorafenib
* Capecitabine + placebo ("dummy medication" with no active drug)

Participants will continue to receive treatments until there is radiographic or clinical progression of disease, side effects which require them to withdraw, pregnancy, protocol non-compliance or withdrawal of consent. Therefore length of participation will vary for individuals. This study is expected to close 31 March 2013.

This is a multicentre study which will take place across Europe, North and South America, Asia, Australia and South Africa. It is anticipated that approximately 519 participants will be recruited worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Age is >=18 years
* Subject has histologically or cytologically confirmed HER2-negative adenocarcinoma of the breast. HER2 status should be determined by an accredited laboratory
* Subject has locally advanced or metastatic disease; locally advanced disease must not be amenable to resection with curative intent. Must have measurable or non-measurable disease (according to RECIST [Response Evaluation Criteria for Solid Tumors] 1.1)
* All computer tomography (CT; with contrast) and magnetic resonance imaging (MRI) used to document disease must have been done <= 4 weeks before randomization. Bone scans (if clinically indicated) must have been done <= 12 weeks prior to randomization
* Subject must have received up to two prior chemotherapy regimens (adjuvant/neo-adjuvant treatments are considered one regimen), and no more than one prior regimen for advanced and/or metastatic disease. Chemotherapy regimens include both targeted and biologic therapy
* Prior regimens must have included an anthracycline (eg, doxorubicin, epirubicin) and a taxane (eg, paclitaxel, docetaxel), either in combination or in separate regimens, in either the neo-adjuvant/adjuvant or the metastatic setting or both, as either monotherapy or as part of a combination with another agent. Sequential regimens will count as a single regimen; multiple neo-adjuvant / adjuvant regimens will count as a single regimen
* Subjects are either resistant to or have failed prior taxane and anthracycline OR Resistant to or have failed prior taxane AND for whom further anthracycline therapy is not indicated (for example, intolerance or cumulative doses of doxorubicin or doxorubicin equivalents [for example, epirubicin)
* Subjects who relapse beyond 12 months after the last taxane or anthracycline dose given in the adjuvant, neo-adjuvant, or metastatic setting are eligible. Further therapy with the agent(s) for a subsequent regimen must have been considered and ruled out, for example due to prior toxicity or intolerance, or based on the local standard of practice
* Prior experimental chemotherapy treatment is allowed, provided it is given in combination with at least one drug approved for the treatment of breast cancer (excluding drugs that target VEGF [Vascular Endothelial Growth Factor] or VEGFR [Vascular Endothelial Growth Factor Receptor], eg, bevacizumab, brivanib, sunitinib, vatalinib).
* Prior hormonal therapy for locally advanced or metastatic breast cancer is allowed. Subjects who are refractory to hormonal therapy are allowed.
* Prior neo-adjuvant or adjuvant chemotherapy is allowed.
* Subject must have discontinued prior chemotherapy (including both targeted and biologic therapies), prior therapeutic radiation therapy, or prior hormonal therapy for locally advanced or metastatic disease >= 4 weeks (28 days) before randomization. Start of study treatment is allowed within less than 28 days of the prior therapy provided that 5 half-lives of the prior treatment drug(s) have elapsed
* ECOG (Eastern Cooperative Oncology Group) performance status 0 or 1
* Adequate bone marrow, liver and renal function within 7 days prior to randomization
* All acute toxic effects of any prior treatment have resolved to NCI-CTCAE (National Cancer Institute-Common Terminology Criteria for Adverse Events) v4.0 Grade 1 or less
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to randomization
* Subjects (men and women) of childbearing potential must agree to use adequate contraception beginning at the signing of the ICF (Informed Consent Form) until at least 30 days after the last dose of study drug.
* Subject must be able to swallow and retain oral medication

Exclusion Criteria:

* HER2 positive breast cancer
* Unknown hormone receptor status (estrogen and progesterone receptor).
* Subjects with bilateral breast cancer or a history of two distinct breast cancers.
* Subjects with inflammatory breast carcinoma.
* Subjects who have received no prior taxane and anthracycline for the treatment of breast cancer (either in adjuvant, neo-adjuvant or metastatic setting).
* Prior use of sorafenib or capecitabine
* Subjects considered by the treating investigator to be appropriate candidates for hormonal therapy as current treatment for locally advanced/metastatic breast cancer
* Subjects with locally advanced disease who are considered by the treating investigator to be appropriate candidates for radiation therapy as current treatment for locally advanced breast cancer
* Subjects with active brain metastases or leptomeningeal disease.
* Subjects with seizure disorder requiring medication.
* Radiation to any lesions <= 4 weeks prior to randomization. Palliative radiation to bone metastasis for pain control is permitted with provisions
* Major surgery, open biopsy, or significant traumatic injury <= 4 weeks
* Evidence or history of bleeding diathesis or coagulopathy. Uncontrolled hypertension, active or clinically significant cardiac disease. Subject with thrombotic, embolic, venus or arterial events
* Subjects with any hemorrhage/bleeding event of NCI-CTCAE v4.0 Grade 3 or higher within 4 weeks before randomization
* Subjects with an infection of NCI-CTCAE v4.0 > Grade 2
* Subjects with a history of human immunodeficiency virus infection or current chronic or active hepatitis B or C infection.
* Subjects who have used strong CYP3A4 inducers (eg, phenytoin, carbamazepine, phenobarbital, St. John's Wort [Hypericum perforatum], dexamethasone at a dose of greater than 16 mg daily, or rifampin [rifampicin], and/or rifabutin) within 28 days before randomization.
* Subjects with any previously untreated or concurrent cancer that is distinct in primary site or histology from breast cancer
* Subjects with a history DHPD (Dihydropyrimidine dehydrogenase) reaction to fluropyrimidine or history of known or suspected allergy or hypersensitivity to any of the study drugs
* Presence of a non-healing wound, non-healing ulcer, or bone fracture
* Women pregnant or breast feeding
* Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 537 (Actual)
Dates: Start 2011-02-21 (Actual); Primary Completion 2014-05-12 (Actual); Study Completion 2017-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (127):
- United States (18):
  - Greenbrae, California
  - Sylmar, California
  - West Palm Beach, Florida
  - Joliet, Illinois
  - Evansville, Indiana
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Jackson, Mississippi
  - Springfield, Missouri
  - Albuquerque, New Mexico
  - Lake Success, New York
  - Durham, North Carolina
  - Philadelphia, Pennsylvania
  - Bristol, Tennessee
  - Memphis, Tennessee
  - El Paso, Texas
  - Burlington, Vermont
  - Madison, Wisconsin
- Argentina (2):
  - Mar del Plata, Buenos Aires
  - Buenos Aires, Ciudad Auton. de Buenos Aires
- Australia (7):
  - Garran, Australian Capital Territory
  - Liverpool, New South Wales
  - Waratah, New South Wales
  - Adelaide, South Australia
  - Bendigo, Victoria
  - Frankston, Victoria
  - Perth, Western Australia
- Austria (2):
  - Linz, Upper Austria
  - Vienna
- Belgium (5):
  - Liège, Liège
  - Bruges
  - Bruxelles - Brussel
  - Edegem
  - Hasselt
- Montreal, Quebec, Canada
- China (6):
  - Shenyang, Liaoning
  - Beijing
  - Nanning
  - Shanghai
  - Tianjin
  - Xi'an
- Czechia (5):
  - České Budějovice
  - Nová Ves pod Pleší
  - Nymburk
  - Olomouc
  - Prague
- France (5):
  - Clermont-Ferrand
  - Lille
  - Nantes
  - Saint-Cloud
  - Toulouse
- Germany (8):
  - Erlangen, Bavaria
  - Frankfurt am Main, Hesse
  - Offenbach, Hesse
  - Cologne, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Leipzig, Saxony
  - Stendal, Saxony-Anhalt
  - Berlin
- Greece (5):
  - Athens
  - Heraklion
  - Ioannina
  - Larissa
  - Pátrai
- Hungary (5):
  - Budapest
  - Nyíregyháza
  - Pécs
  - Szentes
  - Szolnok
- Ireland (3):
  - Cork
  - Dublin
  - Galway
- Israel (5):
  - Beersheba
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Ramat Gan
- Italy (11):
  - Bologna, Emilia-Romagna
  - Forlì-Cesena, Emilia-Romagna
  - Modena, Emilia-Romagna
  - Ravenna, Emilia-Romagna
  - Rome, Lazio
  - Cremona, Lombardy
  - Milan, Lombardy
  - Monza-Brianza, Lombardy
  - Palermo, Sicily
  - Ancona, The Marches
  - Pisa, Tuscany
- Japan (11):
  - Nagoya, Aichi-ken
  - Matsuyama, Ehime
  - Suita, Osaka
  - Hidaka, Saitama
  - Kita-Adachigun, Saitama
  - Bunkyo, Tokyo
  - Koto-ku, Tokyo
  - Chiba
  - Fukuoka
  - Kagoshima
  - Osaka
- Poland (3):
  - Gdansk
  - Gdynia
  - Poznan
- San Juan, Puerto Rico
- Russia (2):
  - Chelyabinsk
  - Kazan'
- South Africa (3):
  - Port Elizabeth, Eastern Cape
  - Johannesburg, Gauteng
  - Pretoria, Gauteng
- Spain (13):
  - Santiago de Compostela, A Coruña
  - Sabadell, Barcelona
  - Terrassa, Barcelona
  - Castellon, Castellón
  - Palma de Mallorca, Illes Baleares
  - Reus, Tarragona
  - A Coruña
  - Barcelona
  - Lleida
  - Madrid
  - Palma de Mallorca
  - Seville
  - Valencia
- Stockholm, Sweden
- United Kingdom (5):
  - Truro, Cornwall
  - Nottingham, Nottinghamshire
  - London
  - Manchester
  - Northwood

REFERENCES:
- [Result] Baselga J, Costa F, Gomez H, Hudis CA, Rapoport B, Roche H, Schwartzberg LS, Petrenciuc O, Shan M, Gradishar WJ. A phase 3 tRial comparing capecitabinE in combination with SorafenIb or pLacebo for treatment of locally advanced or metastatIc HER2-Negative breast CancEr (the RESILIENCE study): study protocol for a randomized controlled trial. Trials. 2013 Jul 22;14:228. doi: 10.1186/1745-6215-14-228. PMID 23876062
- [Result] Baselga J, Zamagni C, Gomez P, Bermejo B, Nagai SE, Melichar B, Chan A, Mangel L, Bergh J, Costa F, Gomez HL, Gradishar WJ, Hudis CA, Rapoport BL, Roche H, Maeda P, Huang L, Meinhardt G, Zhang J, Schwartzberg LS. RESILIENCE: Phase III Randomized, Double-Blind Trial Comparing Sorafenib With Capecitabine Versus Placebo With Capecitabine in Locally Advanced or Metastatic HER2-Negative Breast Cancer. Clin Breast Cancer. 2017 Dec;17(8):585-594.e4. doi: 10.1016/j.clbc.2017.05.006. Epub 2017 May 22. PMID 28830796
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At 154 sites in 22 countries, participants with histologically or cytologically confirmed human epidermal growth factor receptor 2 (HER2)-negative adenocarcinoma of the breast, and locally advanced or metastatic disease, were screened.
Pre-assignment Details: Of 707 participants screened, 537 participants were randomized and 527 participants received at least 1 dose of study treatment. The reasons for 170 screen failures were adverse event in 21 participants, disease progression, recurrence or relapse in 2, consent withdrawn in 16, death in 4, and protocol violation in 127 participants.
Groups:
- Sorafenib (Nexavar, BAY43-9006) + Capecitabine: Sorafenib tablets were administered orally continuously at a total daily dose of 600 mg (200 mg in the morning, 400 mg in the evening) in a 3-week cycle. Capecitabine was administered orally at a total daily dose of 2,000 mg/m^2 (1,000 mg/m^2 twice daily, 12 hours apart). If tolerability criteria were met for a participant, capecitabine dose was escalated to 2,500 mg/m^2 total daily dose (1,250 mg/m^2 twice daily) and sorafenib dose to a total daily dose of 800 mg for that participant.
- Placebo + Capecitabine: Placebo tablets matching with sorafenib were administered orally continuously (1 tablet in the morning, 2 tablets in the evening) in a 3-week cycle. Capecitabine was administered orally at a total daily dose of 2,000 mg/m^2 (1,000 mg/m^2 twice daily, 12 hours apart). If tolerability criteria were met for a participant, capecitabine dose was escalated to 2,500 mg/m^2 total daily dose (1,250 mg/m^2 twice daily) and placebo dose to a total daily dose of 4 tablets (2 tablets twice daily) for that participant.
Period: Overall Study
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Capecitabine | Placebo + Capecitabine
Started | 266 | 271
Participants Received Treatment | 260 | 267
Completed | 0 | 0
Not Completed | 266 | 271
Not completed — Adverse Event | 58 | 21
Not completed — Disease progression/recurrence/relapse | 181 | 223
Not completed — Investi. decision not protocol driven | 5 | 6
Not completed — Non-compliant with study medication | 3 | 2
Not completed — Randomized but not treated | 6 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 2 | 3
Not completed — Withdrawal by Subject | 11 | 9
Not completed — Death | 0 | 1
Not completed — Switch to commercial drug | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Capecitabine | Placebo + Capecitabine | Total
Number analyzed (Participants) | 266 | 271 | 537
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (10.2) | 54.4 (10.9) | 53.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 265 | 268 | 533
  Male | 1 | 3 | 4
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 205 | 212 | 417
  Black | 7 | 4 | 11
  Asian | 50 | 50 | 100
  Hispanic | 4 | 5 | 9
Region of Enrollment [Number; unit: Participants] — Other countries in the below category included Argentina, Australia, China, Israel and Japan.
  Participants
    Europe | 166 | 168 | 334
    North America | 23 | 26 | 49
    Other | 77 | 77 | 154
Eastern Cooperative Oncology Group (ECOG) [Count of Participants; unit: Participants] — ECOG status 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory, able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2=Ambulatory, capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; 3=Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4=Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
  Participants
    ECOG status=0 | 152 | 161 | 313
    ECOG status=1 | 114 | 110 | 224
    ECOG status=2 | 0 | 0 | 0
    ECOG status=3 | 0 | 0 | 0
    ECOG status=4 | 0 | 0 | 0
Number of Prior Chemotherapies for Metastatic Disease [Count of Participants; unit: Participants] — Assessed by Interactive voice response system (IVRS). Participants with more than 1 actual number of prior chemotherapies were combined with participants with 1 prior chemotherapy.
  Participants
    Prior chemotherapies=0 | 114 | 118 | 232
    Prior chemotherapies=1 | 152 | 153 | 305
Hormone Receptor Status [Count of Participants; unit: Participants] — The hormone receptor status was assessed by IVRS, and considered as follows: in case, the tumor expressed estrogen and/or progesterone receptor, the participant was considered to have positive hormone receptor status. Otherwise, if both receptors were not expressed, then participant was considered to have a negative hormone receptor status.
  Participants
    Negative | 83 | 84 | 167
    Positive | 183 | 187 | 370
Visceral Disease at Baseline [Count of Participants; unit: Participants]
  Missing | 1 | 1 | 2
  No | 66 | 57 | 123
  Yes | 199 | 213 | 412

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Assessed by the Independent Review Panel According to Response Evaluation Criteria for Solid Tumors (RECIST) 1.1
Description: PFS was defined as the time from date of randomization to disease progression, radiological or death due to any cause, whichever occurs first. Per RECIST version 1.1, progressive disease was determined when there was at least 20% increase in the sum of diameters of the target lesions, taking as a reference the smallest sum on study (this included the baseline sum if that was the smallest sum on trial). In addition to a relative increase of 20%, the sum had demonstrated an absolute increase of at least 5 mm. Appearance of new lesions and unequivocal progression of existing non-target lesions was also interpreted as progressive disease. Participants without progression or death at the time of analysis were censored at their last date of evaluable tumor evaluation. Median and other 95% confidence intervals (CIs) computed using Kaplan-Meier estimates.
Time Frame: From randomization of the first participant until approximately 3 years or until disease radiological progression
Population: Full Analysis Set (FAS), also considered as Intent-to-treat (ITT) set, was defined as all randomized participants even if randomized but received no drug or if randomized and initially received incorrect drug prior to switching to correct study drug, these were included in FAS.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Capecitabine | Placebo + Capecitabine
Number analyzed (Participants) | 266 | 271
days | 166 [131 to 206] | 165 [126 to 204]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + Capecitabine vs Placebo + Capecitabine; PFS was compared using a stratified log-rank test with a one-sided alpha of 0.005, stratified by region, hormone receptor status, number of previous chemotherapies for metastatic disease. The hazard ratio (sorafenib + capecitabine / placebo + capecitabine) and its 95 percent (%) CIs were calculated using the Cox model, stratified by the above factors. A Hazard ratio of less than (<) 1 indicates superiority of Sorafenib + Capecitabine over Placebo + Capecitabine; Test type: Superiority or Other; p = 0.405618, Log Rank — One-sided p-value from log rank test (stratified per randomization as in interactive voice response system [IVRS]); Hazard Ratio (HR) = 0.973, 95% CI 2-sided [0.779 to 1.217]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from date of randomization to death due to any cause. Participants still alive at the time of analysis were censored at their last known alive date. Median and other 95% CIs computed using Kaplan-Meier estimates.
Time Frame: From randomization of the first participant until approximately 3 years later
Population: FAS
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Capecitabine | Placebo + Capecitabine
Number analyzed (Participants) | 266 | 271
days | 575 [467 to 645] | 616 [546 to 687]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + Capecitabine vs Placebo + Capecitabine; At the time of PFS final analysis, it was OS interim analysis (IA) with 285 total death events. According to protocol specified O'Brien-Fleming type alpha spending function and 285 death events at IA, the prespecified alpha for this analysis was 0.0075 (one-sided). A Hazard ratio < 1 indicates superiority of Sorafenib+Capecitabine over Placebo+Capecitabine; Test type: Superiority or Other; p = 0.930088, Log Rank — One-sided p-value from log rank test (stratified per randomization as in IVRS). OS was compared using a stratified log-rank test, stratified by region, hormone receptor status, number of previous chemotherapies for metastatic disease; Hazard Ratio (HR) = 1.195, 95% CI 2-sided [0.943 to 1.513] — The hazard ratio (sorafenib + capecitabine / placebo + capecitabine) and its 95% CIs were calculated using the Cox model, stratified by randomization factors

3. Secondary Outcome: Time to Progression (TTP) by Central Review
Description: TTP was defined as the time from date of randomization to disease radiological progression by central review. Per RECIST version 1.1, progressive disease was determined when there was at least 20% increase in the sum of diameters of the target lesions, taking as a reference the smallest sum on study (this included the baseline sum if that was the smallest sum on trial). In addition to a relative increase of 20%, the sum had demonstrated an absolute increase of at least 5 mm. Appearance of new lesions and unequivocal progression of existing non-target lesions was also interpreted as progressive disease. Participants without progression or death at the time of analysis were censored at their last date of evaluable tumor evaluation. Median and other 95% confidence intervals (CIs) computed using Kaplan-Meier estimates.
Time Frame: From randomization of the first participant until approximately 3 years later or until disease radiological progression
Population: FAS
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Capecitabine | Placebo + Capecitabine
Number analyzed (Participants) | 266 | 271
days | 168 [139 to 215] | 165 [127 to 208]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + Capecitabine vs Placebo + Capecitabine; TTP was compared using a stratified log-rank test with a one-sided alpha of 0.025, stratified by region, hormone receptor status, number of previous chemotherapies for metastatic disease. A Hazard ratio <1 indicates superiority of Sorafenib+Capecitabine over Placebo+Capecitabine; Test type: Superiority or Other; p = 0.2105, Log Rank — One-sided p-value from log rank test (stratified per randomization as in IVRS); Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.723 to 1.146] — The hazard ratio (sorafenib + capecitabine / placebo + capecitabine) and its 95% CIs were calculated using the Cox model, stratified by the above factors

4. Secondary Outcome: Objective Response Rate (ORR) by Central Review
Description: ORR was defined as the best tumor response (Complete Response [CR] or Partial Response [PR]) observed during treatment or within 30 days after termination of study treatment, assessed according to the RECIST version 1.1. CR=all target lesions disappeared, and any pathological lymph node, whether target or non-target, had a reduction in short axis to <10 mm. If any residual lesion was present, cyto-histology was made available to unequivocally document benignity. PR=at least 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. ORR=CR+PR. CR and PR were confirmed by another scan at least 4 weeks later.
Time Frame: From randomization of the first participant until approximately 3 years later or until disease radiological progression
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage (%) of participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Capecitabine | Placebo + Capecitabine
Number analyzed (Participants) | 266 | 271
Percentage (%) of participants | 13.5 [9.7 to 18.2] | 15.5 [11.4 to 20.4]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + Capecitabine vs Placebo + Capecitabine; ORR and 95% CI based on Cochran Mantel-Haenszel Test stratified by region, hormone receptor status, number of previous chemotherapies for metastatic disease. Difference = (Placebo + Capecitabine) - (Sorafenib + Capecitabine); Test type: Superiority or Other; p = 0.257412, Cochran-Mantel-Haenszel — One-sided p-value from Cochran Mantel-Haenszel test (stratified per randomization as in IVRS); Percent Difference = 1.93, 95% CI 2-sided [-3.9 to 7.77]

5. Secondary Outcome: Disease Control Rate (DCR) by Central Review
Description: DCR was defined as the proportion of participants whose best response was CR, PR, stable disease (SD) or Non-CR/Non-PD. Per RECIST version 1.1, CR=all target lesions disappeared, any pathological lymph node, target/non-target, a reduction in short axis to <10 mm. PR=at least 30% decrease in the sum of diameters of target lesions taking as reference baseline sum diameters. PD=at least 20% increase in the sum of diameters of the target lesions, taking as a reference smallest sum on study. Appearance of new lesions and unequivocal progression of existing non-target lesions. SD=neither sufficient shrinkage qualified for PR nor sufficient increase qualified for PD, taking smallest sum of diameters as a reference. Non-CR/Non-PD=persistence of 1/more non-target lesion(s) and/or maintenance of tumor marker level above normal limits. DCR=CR+PR+SD or Non-CR/Non-PD. CR and PR confirmed by another scan at least 4 weeks later. SD and Non-CR/Non-PD documented at least 6 weeks after randomization.
Time Frame: From randomization of the first participant until approximately 3 years later or until disease radiological progression
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage (%) of participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Capecitabine | Placebo + Capecitabine
Number analyzed (Participants) | 266 | 271
percentage (%) of participants | 60.5 [54.4 to 66.4] | 58.3 [52.2 to 64.2]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + Capecitabine vs Placebo + Capecitabine; DCR and 95% CI based on "general association Cochran-Mantel-Haenszel statistic" with one-sided alpha of 0.025 stratified by number of prior chemotherapies for metastatic disease, hormone receptor status, and region. Difference = Placebo + Capecitabine - Sorafenib + Capecitabine; Test type: Superiority or Other; p = 0.284674, Cochran-Mantel-Haenszel — One-sided p-value from Cochran-Mantel-Haenszel test (stratified per randomization as in IVRS); Percent Difference = -2.34, 95% CI 2-sided [-10.4 to 5.72]

6. Secondary Outcome: Duration of Response (DOR) by Central Reader
Description: DOR was defined as the time from date of first response (CR or PR) to the date when PD is first documented, or to the date of death, whichever occurred first according to RECIST version 1.1. CR=all target lesions disappeared, and any pathological lymph node, whether target or non-target, had a reduction in short axis to <10 mm. If any residual lesion was present, cyto-histology was made available to unequivocally document benignity. PR=at least 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Participants still having CR or PR and have not died at the time of analysis were censored at their last date of tumor evaluation. DOR defined for confirmed responders only (that is, CR or PR). 'NA' indicates that value could not be estimated due to censored data. Median and 95% CIs were computed using Kaplan-Meier estimates.
Time Frame: From randomization of the first participant until approximately 3 years later or until disease radiological progression
Population: Only responders in FAS were evaluated for this outcome measure.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Capecitabine | Placebo + Capecitabine
Number analyzed (Participants) | 36 | 42
days | 313 [209 to NA] — Value could not be estimated due to censored data. | 290 [169 to NA] — Value could not be estimated due to censored data.

7. Other Pre Specified Outcome: Patient Reported Outcomes: Functional Assessment of Cancer Therapy-Breast Symptom Index (8 Item) (FBSI-8)
Description: The FBSI-8 was an 8-item questionnaire. Participants responded to each item using a 5-point Likert-type scale ranging from 0 (not at all) to 4 (very much). A total scale score was calculated (range from 0 to 32), with higher scores indicating low symptomatology and reflecting a better Health-Related Quality of Life (HRQoL). The results on the analysis of covariance (ANCOVA) of time-adjusted area under curve (AUC) for the FBSI-8 score were reported. The time-adjusted AUC was calculated by dividing the AUC by duration (in days) over the period of interest, and reported as 'scores on a scale'.
Time Frame: Day 1 of Cycles 1, 3, 5, 7, 9, 11, 13, 16, 19, 22, 25, 28, 31, 34, 37, and end of treatment (EOT, 21 days after last dose of study drug)
Population: FAS participants with a baseline assessment and at least one post-baseline assessment during the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Capecitabine | Placebo + Capecitabine
Number analyzed (Participants) | 233 | 243
Scores on a scale | 20.915 [20.459 to 21.37] | 21.356 [20.911 to 21.801]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + Capecitabine vs Placebo + Capecitabine; Estimate of Difference (least squares mean [LSM] difference) = (Sorafenib + Capecitabine) - (Placebo + Capecitabine). The difference between the two treatment groups was evaluated with an analysis of covariance model using the baseline score and the same stratification factors as used for randomization (IVRS) as covariates; Test type: Superiority or Other; LSM Difference = -0.441, 95% CI 2-sided [-0.967 to 0.086]

8. Other Pre Specified Outcome: Patient Reported Outcomes: Euroqol-5 Dimensions (EQ-5D) - Index Score
Description: The EQ-5D was a generic Quality of life (QoL) based instrument validated in cancer populations. EQ-5D questionnaire contained a 5-item descriptive system of health states (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and visual analogue scale (VAS). A single HRQoL score ranging from -0.59 to 1 was generated from standard scoring algorithm developed by the EuroQoL was the EQ-5D index score, higher scores represent better health status. A change of at least 0.10 to 0.12 points was considered clinically meaningful. The results on the ANCOVA of time-adjusted AUC for the EQ-5D - Index Score were reported. The time-adjusted AUC was calculated by dividing the AUC by duration (in days) over the period of interest, and reported as 'scores on a scale'.
Time Frame: Day 1 of Cycles 1, 3, 5, 7, 9, 11, 13, 16, 19, 22, 25, 28, and EOT (21 days after last dose of study drug)
Population: FAS participants with a baseline assessment and at least one post-baseline assessment during the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Capecitabine | Placebo + Capecitabine
Number analyzed (Participants) | 236 | 247
Scores on a scale | 0.665 [0.641 to 0.688] | 0.69 [0.667 to 0.713]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + Capecitabine vs Placebo + Capecitabine; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; LSM Difference = -0.025, 95% CI 2-sided [-0.053 to 0.002]

9. Other Pre Specified Outcome: Patient Reported Outcomes: Euroqol-5 Dimensions (EQ-5D) - Visual Analogue Scale (VAS) Score
Description: The EQ-5D was a generic QoL preference based instrument and has been validated in the cancer populations. VAS was generated from 0 (worst imaginable health state) to 100 (best imaginable health state). This VAS score was referred to as the EQ-5D self-reported health status score. The results on ANCOVA of time-adjusted AUC were reported. The time-adjusted AUC was calculated by dividing the AUC by duration (in days) over the period of interest, and reported as 'scores on a scale'.
Time Frame: Day 1 of Cycles 1, 3, 5, 7, 9, 11, 13, 16, 19, 22, 25, 28, and EOT (21 days after last dose of study drug)
Population: FAS participants with a baseline assessment and at least one post-baseline assessment during the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Capecitabine | Placebo + Capecitabine
Number analyzed (Participants) | 235 | 244
Scores on a scale | 67.532 [65.87 to 69.19] | 69.228 [67.6 to 70.86]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + Capecitabine vs Placebo + Capecitabine; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; LSM Difference = -1.696, 95% CI 2-sided [-3.619 to 0.227]

10. Other Pre Specified Outcome: Maximum Observed Drug Concentration (Cmax) of Capecitabine and 5-fluorouracil
Description: Maximum observed drug concentration, directly taken from analytical data. Geometric mean and percentage geometric coefficient of variation (%CV) were reported. In the listed categories below, 'N' signifies the number of evaluable participants for the drug administered.
Time Frame: Pre-dose and 0.5, 1, 2, and 4 hours after capecitabine dosing at Cycle 2, Day 14
Population: Pharmacokinetic Analysis Set (PKS) included all participants with a valid pharmacokinetic profile of capecitabine.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram per liter
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Capecitabine | Placebo + Capecitabine
Number analyzed (Participants) | 56 | 84
milligram per liter
  Capecitabine | 6.05 (79) | 4.68 (72)
  5-fluorouracil: number analyzed (Participants) | 51 | 84
  5-fluorouracil | 0.434 (105) | 0.382 (67)
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + Capecitabine vs Placebo + Capecitabine; Statistical analysis for Cmax: 5-fluorouracil; Test type: Superiority or Other; Ratio of geometric least square means = 1.14, 90% CI 2-sided [0.92 to 1.40]
Statistical Analysis 2: Comparison: Sorafenib (Nexavar, BAY43-9006) + Capecitabine vs Placebo + Capecitabine; Statistical analysis for Cmax: Capecitabine; Test type: Superiority or Other; Ratio of geometric least square means = 1.29, 90% CI 2-sided [1.07 to 1.56]

11. Other Pre Specified Outcome: Area Under Curve From Time Zero to Last Quantifiable Concentration (AUC[0-tlast]) of Capecitabine and 5-fluorouracil
Description: AUC(0-tlast) is defined as AUC from time 0 to the last data point, calculated up by linear trapezoidal rule, down by logarithmic trapezoidal rule. Geometric mean and percentage geometric coefficient of variation (%CV) were reported. In the listed categories below, 'N' signifies the number of evaluable participants for the drug administered.
Time Frame: Pre-dose and 0.5, 1, 2, and 4 hours after capecitabine dosing at Cycle 2, Day 14
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram*hour per liter
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Capecitabine | Placebo + Capecitabine
Number analyzed (Participants) | 56 | 84
milligram*hour per liter
  Capecitabine | 7.12 (50) | 5.13 (48)
  5-fluorouracil: number analyzed (Participants) | 51 | 84
  5-fluorouracil | 0.621 (71) | 0.557 (47)
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + Capecitabine vs Placebo + Capecitabine; Statistical analysis for AUC(0-tlast): 5-fluorouracil; Test type: Superiority or Other; Ratio of geometric least square means = 1.11, 90% CI 2-sided [0.95 to 1.30]
Statistical Analysis 2: Comparison: Sorafenib (Nexavar, BAY43-9006) + Capecitabine vs Placebo + Capecitabine; Statistical analysis for AUC(0-tlast): Capecitabine; Test type: Superiority or Other; Ratio of geometric least square means = 1.39, 90% CI 2-sided [1.22 to 1.58]

12. Other Pre Specified Outcome: Number of Participants With Treatment-emergent Grade 3 and 4 Laboratory Abnormalities
Description: Hematological (anemia, hemoglobin, international normalized ratio [INR], lymphocyte, neutrophil, platelet, white blood cell [WBC]), biochemical (ALT [alanine aminotransferase], AST [aspartate aminotransferase], GGT [gamma-glutamyl-transferase], lipase, hypoalbuminemia, hypocalcemia, hyperglycemia, hyperuricemia) evaluations were done. Common terminology criteria for adverse events (CTCAE) version 4-Grade 3: Severe or medically significant; hospitalization or prolongation of hospitalization and CTCAE version 4-Grade 4: life-threatening consequences; urgent intervention were indicated.
Time Frame: From the start of study treatment up to 30 days after the last dose
Population: Safety Analysis Set (SAF) was comprised of all randomized participants who received at least one dose of study medication (sorafenib, placebo or capecitabine). Participants were analyzed as treated.
Measure: Number; unit: Participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Capecitabine | Placebo + Capecitabine
Number analyzed (Participants) | 260 | 267
Participants
  Anemia (grade 3) | 12 | 7
  Hemoglobin increased (grade 3) | 0 | 3
  INR increased (grade 3) | 9 | 9
  Lymphocyte count decreased (grade 3) | 20 | 17
  Neutrophil count decreased (grade 3) | 11 | 19
  Platelet count decreased (grade 3) | 6 | 2
  WBC decreased (grade 3) | 15 | 13
  ALT increased (grade 3) | 4 | 5
  AST increased (grade 3) | 10 | 5
  Alkaline phosphatase increased (grade 3) | 12 | 13
  Bilirubin increased (grade 3) | 9 | 1
  GGT increased (grade 3) | 22 | 21
  Lipase increased (grade 3) | 19 | 12
  Serum amylase increased (grade 3) | 8 | 4
  Hypoalbuminemia (grade 3) | 4 | 2
  Hypocalcemia (grade 3) | 9 | 6
  Hypokalemia (grade 3) | 20 | 11
  Hyponatremia (grade 3) | 9 | 7
  Hypophosphatemia (grade 3) | 47 | 15
  Hyperglycemia (grade 3) | 9 | 10
  Lymphocyte count decreased (grade 4) | 3 | 2
  Neutrophil count decreased (grade 4) | 7 | 7
  Platelet count decreased (grade 4) | 1 | 7
  WBC decreased (grade 4) | 2 | 3
  ALT increased (grade 4) | 3 | 0
  GGT increased (grade 4) | 6 | 2
  Lipase increased (grade 4) | 5 | 1
  Hypokalemia (grade 4) | 2 | 4
  Hyponatremia (grade 4) | 4 | 0
  Hypophosphatemia (grade 4) | 5 | 0
  Hyperuricemia (grade 4) | 5 | 0

ADVERSE EVENTS:
Time Frame: From start of study drug administration until 30 days after the last dose of study medication intake.
Groups:
- Sorafenib (Nexavar, BAY43-9006) + Capecitabine: Sorafenib tablets were administered orally continuously at a total daily dose of 600 mg (200 mg in the morning, 400 mg in the evening) in a 3-week cycle. Capecitabine was administered orally at a total daily dose of 2,000 mg/m^2 (1,000 mg/m^2 twice daily, 12 hours apart). If tolerability criteria were met for a subject, capecitabine dose was escalated to 2,500 mg/m^2 total daily dose (1,250 mg/m^2 twice daily) and sorafenib dose to a total daily dose of 800 mg for that subject.
- Placebo + Capecitabine: Placebo tablets matching with sorafenib were administered orally continuously (1 tablet in the morning, 2 tablets in the evening) in a 3-week cycle. Capecitabine was administered orally at a total daily dose of 2,000 mg/m^2 (1,000 mg/m^2 twice daily, 12 hours apart). If tolerability criteria were met for a subject, capecitabine dose was escalated to 2,500 mg/m^2 total daily dose (1,250 mg/m^2 twice daily) and placebo dose to a total daily dose of 4 tablets (2 tablets twice daily) for that subject.
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + Capecitabine | Placebo + Capecitabine
Serious Adverse Events (participants affected / at risk) | 80/260 | 71/267
Other Adverse Events (participants affected / at risk) | 256/260 | 248/267
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) + Capecitabine (N=260) | Placebo + Capecitabine (N=267)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 5 (6)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Aplasia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Eye symptom (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Acute abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (2) | 2 (7)
Colitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 8 (8)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (7) | 1 (1)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neutropenic colitis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Death (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 2 (2) | 2 (2)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (3)
General physical health deterioration (General disorders) | 3 (3) | 3 (3)
Gallbladder pain (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Cytomegalovirus enterocolitis (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Biopsy lung (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Central nervous system mass (Nervous system disorders) | 0 (0) | 1 (1)
Cytotoxic oedema (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 3 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 11 (11)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Pulmonary microemboli (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Tracheal obstruction extrinsic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Pleurodesis (Surgical and medical procedures) | 2 (2) | 0 (0)
Central venous catheterisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Hepatectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Axillary lymphadenectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Cancer surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 3 (3)
Peripheral artery occlusion (Vascular disorders) | 1 (3) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) + Capecitabine (N=260) | Placebo + Capecitabine (N=267)
Anaemia (Blood and lymphatic system disorders) | 31 (37) | 32 (37)
Neutropenia (Blood and lymphatic system disorders) | 12 (22) | 24 (46)
Lacrimation increased (Eye disorders) | 0 (0) | 16 (21)
Abdominal pain (Gastrointestinal disorders) | 33 (40) | 28 (41)
Abdominal pain upper (Gastrointestinal disorders) | 35 (44) | 19 (22)
Constipation (Gastrointestinal disorders) | 53 (67) | 33 (36)
Diarrhoea (Gastrointestinal disorders) | 123 (291) | 98 (190)
Dyspepsia (Gastrointestinal disorders) | 16 (19) | 25 (31)
Nausea (Gastrointestinal disorders) | 101 (166) | 97 (150)
Stomatitis (Gastrointestinal disorders) | 45 (54) | 24 (29)
Vomiting (Gastrointestinal disorders) | 65 (118) | 53 (83)
Asthenia (General disorders) | 49 (67) | 51 (69)
Fatigue (General disorders) | 79 (101) | 81 (102)
Influenza like illness (General disorders) | 5 (9) | 15 (19)
Mucosal inflammation (General disorders) | 39 (49) | 19 (20)
Oedema peripheral (General disorders) | 9 (10) | 23 (29)
Pyrexia (General disorders) | 28 (31) | 32 (39)
Nasopharyngitis (Infections and infestations) | 24 (35) | 23 (28)
Upper respiratory tract infection (Infections and infestations) | 15 (15) | 11 (12)
Urinary tract infection (Infections and infestations) | 16 (21) | 15 (16)
Alanine aminotransferase increased (Investigations) | 27 (34) | 21 (24)
Aspartate aminotransferase increased (Investigations) | 27 (32) | 23 (26)
Blood bilirubin increased (Investigations) | 19 (27) | 17 (26)
Gamma-glutamyltransferase increased (Investigations) | 14 (14) | 4 (4)
Lipase increased (Investigations) | 13 (15) | 5 (5)
Neutrophil count decreased (Investigations) | 14 (27) | 10 (22)
Weight decreased (Investigations) | 28 (28) | 12 (13)
White blood cell count decreased (Investigations) | 17 (23) | 12 (23)
Hypokalaemia (Metabolism and nutrition disorders) | 22 (24) | 15 (19)
Hypophosphataemia (Metabolism and nutrition disorders) | 16 (22) | 4 (5)
Decreased appetite (Metabolism and nutrition disorders) | 53 (63) | 38 (40)
Arthralgia (Musculoskeletal and connective tissue disorders) | 35 (54) | 27 (33)
Back pain (Musculoskeletal and connective tissue disorders) | 33 (39) | 33 (34)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 17 (24) | 6 (6)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 17 (21)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 (32) | 21 (28)
Dizziness (Nervous system disorders) | 21 (26) | 22 (26)
Dysgeusia (Nervous system disorders) | 12 (13) | 20 (20)
Headache (Nervous system disorders) | 35 (49) | 36 (45)
Anxiety (Psychiatric disorders) | 19 (19) | 12 (12)
Insomnia (Psychiatric disorders) | 16 (16) | 12 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (25) | 23 (25)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 32 (34) | 41 (47)
Alopecia (Skin and subcutaneous tissue disorders) | 44 (49) | 6 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 19 (23) | 17 (19)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 206 (288) | 158 (228)
Rash (Skin and subcutaneous tissue disorders) | 48 (58) | 22 (29)
Hypertension (Vascular disorders) | 69 (92) | 16 (21)

LIMITATIONS AND CAVEATS:
Results of exploratory analysis of biomarkers are anticipated in the month of February, 2016.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bayer will have up to 30/45 days to review publications, and may request an additional publication delay of up to 60 days to allow for filing a Patent Application (if applicable).

No publication of single center data should be done prior to publication of multi-center data.